CLINICAL TRIAL: NCT07181928
Title: Is Mentalization-based Therapy More Effective for Adolescents With Disruptive and Dissocial Disorders Than TAU-plus (Emotion-focused Parent Training With Supportive Child Psychiatric Care)?
Brief Title: Is Mentalization-based Therapy More Effective Than Treatment-as-usual for Adolescents With Dissocial Disorders?
Acronym: MEDAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Vereinigung für analytische und tiefenpsychologisch fundierte Kinder- & Jugendlichen- Psychotherapie (Unknown)
Responsible Party: Principal Investigator, Svenja Taubner, Prof. Dr. phil. Svenja Taubner, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tau 2025 1/2
Record Dates: First submitted 2025-08-01; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Conduct Disorders in Adolescence; Oppositional Defiant Disorder
Keywords: Adolescence; MBT; Conduct Disorder; Externalizing behaviour disorders; Treatment-as-usual
MeSH Terms: conditions — Oppositional Defiant Disorder; Conduct Disorder | interventions — Mentalization-Based Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mentalization-Based Therapy (MBT) (Experimental): 45 adolescents diagnosed with conduct disorder/oppositional defiant disorder will receive MBT over 10 months. The patients have 30 individual sessions weekly conducted by one therapist with formal training in MBT. Additionally, the patient receives 5 sessions together with the parents and the parents will have another 5 sessions without the patient.
  Interventions: Behavioral: Mentalization-Based Therapy (MBT)
- Treatment-as-usual-plus (TAU-plus) (Active Comparator): 45 adolescents diagnosed with conduct disorder/oppositional defiant disorder will receive standard psychiatric care over 10 months and their parents will participate in the Emotion Focused Skills Training (EFST). The patient receives individual psychiatric sessions at least two per quarter depending on the adolescent's needs. The individual sessions are conducted by a child and adolescent psychiatrist and/or by a therapist working under their supervision. EFST includes an intake session, 5 two-hour group sessions (6-12 parents, led by two therapists), and a final individual session.
  Interventions: Behavioral: Treatment-as-usual-plus (TAU-plus)

INTERVENTIONS:
Behavioral: Mentalization-Based Therapy (MBT) — MBT is a manualized psychodynamic therapy based on attachment theory, designed to restore adolescents' mentalizing in general and in emotionally stressful situations and relationships. It targets to rebuilt epistemic trust, to successfully mentalize oneself and others.
  Arms: Mentalization-Based Therapy (MBT)
Behavioral: Treatment-as-usual-plus (TAU-plus) — The adolescents receive supportive child psychiatric consultations. For the parents the EFST sessions combine mindfulness, theoretical input, and experiential practice. Parents learn and apply four core skills: validation, repair, motivation, and setting boundaries.
  Arms: Treatment-as-usual-plus (TAU-plus)

SUMMARY:
The goal of this clinical trial is to investigate if Mentalization-based therapy (MBT) is superior to enhanced usual care (treatment-as-usual-plus (TAU-plus)) for adolescents with disruptive behavior or dissocial disorders.

MBT is an intervention that aims to improve mentalizing. Mentalizing is the ability to reflect on mental states in oneself and others that motivate behavior. TAU-plus consists of psychiatric care for the adolescent, along with additional emotion-focused skills training for the parents.

Participants will be randomized in one of two groups using one study center.

DETAILED DESCRIPTION:
The study includes adolescents between the ages 12 to 19 of any gender who have been diagnosed with Oppositional defiant or Conduct-dissocial disorder (serious problems with following rules or criminal behavior).

The diagnosis is the primary outcome, which is assessed based on a diagnostic interview. Secondary outcomes include antisocial behavior, quality of life, symptom burden, and personality functioning (measured through self-report questionnaires), as well as aggressive behavior (measured through interview).

During the study, there will be monthly process assessments. In these assessments, participants will be asked questions about mentalizing, emotion regulation, therapy experience, antisocial behavior, and how much they trust others. These variables are considered mediators of changes in outcome.

Participants will also be interviewed regarding personality functioning to investigate whether dissocial disorders are related to personality disorders.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Oppositional defiant disorder (ODD) / Conduct-dissocial disorder (CDD) (ICD-11: 6C90-6C91; ICD-10: F91.0-F91.9; DSM-5: 312.81, 313.81)
* Aged 12 to 19 years
* Living with their parents
* Provide written informed consent (plus parental consent for minors)
* At least one parent provides written informed consent and agrees to active participation in treatment and study, including randomization

Exclusion Criteria:

* Severe acute substance dependence requiring inpatient detoxification
* Acute psychotic symptoms or early-onset schizophrenia
* Neurological impairments or intellectual disability (IQ < 80)
* Insufficient proficiency in German
* Other clinical contraindications for outpatient psychotherapy (e.g., acute suicidality)

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Remission rate based on diagnostic criteria for Disruptive behavior or Dissocial disorders | Day 0, Month 14
  Remission is defined as the proportion of participants no longer meeting full diagnostic criteria for Conduct-dissocial disorder (CDD) or Oppositional defiant disorder (ODD). CDD is assessed with the "Diagnostisches Interview bei psychischen Störungen - Version für Jugendlichen" (J-DIPS) and ODD with the "Diagnostisches Interview bei psychischen Störungen im Kindes- und Jugendalter" (K-DIPS).

SECONDARY OUTCOMES:
Aggressive behavior assessed with the german "Modified Overt Aggression Scale" (MOAS-D) | day 0, month 11 month 14
  Score range: 0 - 300, with higher score representing higher value of aggressive behavior
Social aggression assessed with the subscale from Subtypes of Antisocial Behavior Questionnaire (STAB) | day 0 month 11 and month 14
  Score range 11 - 55, with higher score representing higher value of Social aggression
Quality of life assessed with the Kidscreen 10 Index | day 0, month 11, month 14
  Score range: 10-50, with higher scores representing better quality of life
Symptom burden assessed with the Strengths and Difficulties Questionnaire (SDQ) | day 0, month 11, month 14
  Score range: 0 - 40, with higher score representing higher value of difficulties or strengths respectively
Participation assessed with the mini self-rating for psychological activities and participation (Mini-ICF-APP) | day 0, month 14
  Score range: 0 - 7, with higher score represeting higher value of overall capacity level
Gender typicality assessed with the "Instrument zur Erfassung des Geschlechtsrollen-Selbstkonzepts im Jugendalter" (GRI-JUG) | day 0, month 14
  There are four subscales - femenine positive and negative and Masculine positive and negative. Score range for each subscale: 1-5, with high scores indicate a high expression of the respective facet of the gender role self-concept.
Personality functioning assessed with the Level of Personality Functioning Brief Form (LPFS-BF) | day 0, month 11, month 14
  Score range: 12-48, with higher score representing higher value of personality pathology

CONTACTS AND LOCATIONS:
Overall Officials: Svenja Taubner, Prof. Dr., Study Director — Institut für Psychosoziale Prävention, Ruprecht-Karls-Universität Heidelberg
Locations (1):
- Institut für Psychosoziale Prävention, Ruprecht-Karls-Universität Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No
Data is too sensitive

REFERENCES:
- [Background] Korlat S, Holzer J, Schultes MT, Buerger S, Schober B, Spiel C, Kollmayer M. Benefits of Psychological Androgyny in Adolescence: The Role of Gender Role Self-Concept in School-Related Well-Being. Front Psychol. 2022 May 19;13:856758. doi: 10.3389/fpsyg.2022.856758. eCollection 2022. PMID 35664189
- [Background] Kay SR, Wolkenfeld F, Murrill LM. Profiles of aggression among psychiatric patients. I. Nature and prevalence. J Nerv Ment Dis. 1988 Sep;176(9):539-46. doi: 10.1097/00005053-198809000-00007. PMID 3418327
- [Background] Neuschwander M, In-Albon T, Adornetto C, Roth B, Schneider S. [Interrater reliability of the <<Diagnostic Interview bei psychischen Storungen im Kindes- und Jugendalter (Kinder-DIPS)]. Z Kinder Jugendpsychiatr Psychother. 2013 Sep;41(5):319-34. doi: 10.1024/1422-4917//a000247. German. PMID 23988834
- [Background] Spitzer C, Muller S, Kerber A, Hutsebaut J, Brahler E, Zimmermann J. [The German Version of the Level of Personality Functioning Scale-Brief Form 2.0 (LPFS-BF): Latent Structure, Convergent Validity and Norm Values in the General Population]. Psychother Psychosom Med Psychol. 2021 Jul;71(7):284-293. doi: 10.1055/a-1343-2396. Epub 2021 Mar 10. German. PMID 33694153
- [Background] Henning A, Linden M, Muschalla B. Self- and observer ratings of capacity limitations in patients with neurological conditions. Brain Impair. 2023 Dec;24(3):586-600. doi: 10.1017/BrImp.2022.26. Epub 2022 Nov 17. PMID 38167355
- [Background] Klasen H, Woerner W, Rothenberger A, Goodman R. [German version of the Strength and Difficulties Questionnaire (SDQ-German)--overview and evaluation of initial validation and normative results]. Prax Kinderpsychol Kinderpsychiatr. 2003 Sep;52(7):491-502. German. PMID 14526759
- [Background] Ravens-Sieberer U, Herdman M, Devine J, Otto C, Bullinger M, Rose M, Klasen F. The European KIDSCREEN approach to measure quality of life and well-being in children: development, current application, and future advances. Qual Life Res. 2014 Apr;23(3):791-803. doi: 10.1007/s11136-013-0428-3. Epub 2013 May 18. PMID 23686556
- [Background] Burt SA, Donnellan MB. Development and validation of the Subtypes of Antisocial Behavior Questionnaire. Aggress Behav. 2009 Sep-Oct;35(5):376-98. doi: 10.1002/ab.20314. PMID 19618380